CLINICAL TRIAL: NCT04748848
Title: A Phase 1/2, Open-label, Multicenter Dose Escalation and Dose Expansion Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of CC-90011 in Combination With Venetoclax and Azacitidine in R/R Acute Myeloid Leukemia (AML) and Treatment-naïve Subjects With AML Who Are Not Eligible for Intensive Induction Chemotherapy
Brief Title: A Safety, Tolerability and Preliminary Efficacy Study of CC-90011 in Combination With Venetoclax and Azacitidine in R/R Acute Myeloid Leukemia and Treatment-naïve Participants Not Eligible for Intensive Therapy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business objectives have changed.
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CC-90011-AML-002; U1111-1251-6973 (Registry Identifier: WHO); 2020-005341-16 (EudraCT Number)
Record Dates: First submitted 2021-02-02; First posted 2021-02-10 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Leukemia, Myeloid
Keywords: Acute Myeloid Leukemia; CC-90011; Venetoclax; Azacitidine; LSD-1 inhibitor; Minimal residual disease
MeSH Terms: conditions — Leukemia, Myeloid; Leukemia, Myeloid, Acute; Neoplasm, Residual | interventions — pulrodemstat besilate; venetoclax; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CC-90011 in combination with Venetoclax and Azacitidine in Dose Escalation (Experimental): CC-90011 in combination with venetoclax and azacitidine in dose escalation
  Interventions: Drug: CC-90011; Drug: Venetoclax; Drug: Azacitidine
- Venetoclax and Azacitidine (Experimental): Venetoclax and Azacitidine control arm in dose expansion. The participants will be randomized to the treatment arm or control arm at a 2:1 ratio.
  Interventions: Drug: Azacitidine; Drug: Venetoclax
- CC-90011 in combination with Venetoclax and Azacitidine in Dose Expansion (Experimental): CC-90011 in combination with venetoclax and azacitidine in dose expansion
  Interventions: Drug: Venetoclax; Drug: Azacitidine; Drug: CC-90011

INTERVENTIONS:
Drug: CC-90011 — CC-90011 will be given PO on Days 1, 8, and 15 of continuous 4-week (28-day) cycle. The dose escalation is designed to explore three dose levels of CC-90011, for example 20, 40, and 60 mg as determined by Bayesian design.
  Arms: CC-90011 in combination with Venetoclax and Azacitidine in Dose Escalation
Drug: Venetoclax — Venetoclax is administered orally QD on Days 1 to 28 of each 28-day cycle with a brief dose ramp-up for Cycle 1 with the dosing of 100 mg on Day 1, 200 mg on Day 2, and 400 mg on Day 3. Venetoclax should be administered at 400 mg on subsequent days.
  Arms: CC-90011 in combination with Venetoclax and Azacitidine in Dose Escalation; CC-90011 in combination with Venetoclax and Azacitidine in Dose Expansion
Drug: Azacitidine — Azacitidine is administered on Days 1 to 7 of each 28-day cycle as an IV infusion or SC injection at 75 mg/m2
Drug: Venetoclax — Venetoclax is administered orally QD on Days 1 to 28 of each 28-day cycle
  Arms: Venetoclax and Azacitidine
Drug: CC-90011 — CC-90011 will be given PO on Days 1, 8, and 15 of continuous 4-week (28-day) cycle at the recommended phase to dose of CC-90011 confirmed in dose escalation.
  Arms: CC-90011 in combination with Venetoclax and Azacitidine in Dose Expansion

SUMMARY:
CC-90011-AML-002 is a Phase 1/2, open-label, multicenter study to assess the safety, tolerability, and preliminary efficacy of CC-90011 given concurrently with Venetoclax and Azacitidine. This study will include 3 parts: a dose escalation part in R/R AML, a dose escalation part in ndAML (treatment-naïve participants with AML who are ≥ 75 years of age or are ≥ 18 to 74 years of age and otherwise not eligible for intensive induction chemotherapy), and a randomized dose expansion part in ndAML of Venetoclax and Azacitidine with or without CC-90011.

ELIGIBILITY:
Inclusion Criteria:

Participants must satisfy the following criteria to be enrolled in the study:

All participants (Parts I, II, and III):

1. Participant must understand and voluntarily sign an Informed Consent Form (ICF) prior to any study-related assessments/procedures being conducted.

3. Participant must have a projected life expectancy of at least 12 weeks. 4. Participant has Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.

5. Participants must have the required protocol baseline laboratory values 6. Participant has adequate organ function 7. Participant must be able and willing to undergo hospitalization, hydration, and treatment with a uric acid-reducing agent prior to the first dose of venetoclax and during Cycle 1.

Part I only:

8. Relapsed and/or refractory acute myeloid leukemia (AML) as defined by the World Health Organization (WHO) Classification and is ≥ 18 years of age at the time of signing the ICF who are not eligible to receive further intensive therapy and:

1. Has failed to have a complete remission (CR) or CR with incomplete hematologic recovery (Cri) after induction plus reinduction with intensive chemotherapy (anthracycline plus cytarabine containing regimens) or 2 cycles of low intensity therapy (either 2 cycles of the same regimen or 1 cycle of 2 different regimens) OR
2. Has relapsed from CR from either intensive or low-intensity therapy. Participants with second relapse are also eligible

Part II and Part III only:

9. Histologically confirmed treatment naïve Acute myeloid leukemia (AML) as defined by the 2008 World Health Organization (WHO) Classification, including secondary AML and therapy related AML, and is ≥ 75 years of age at the time of signing the ICF, or is ≥ 18 to 74 years at the time of signing the ICF with comorbidities precluding the use of intensive induction chemotherapy 10. Participant has not received prior therapy for AML with the exception of hydroxyurea to treat hyperleukocytosis.

Exclusion Criteria:

The presence of any of the following will exclude a participant from enrollment:

All participants (Parts I, II, and III):

1. Participant is suspected or proven to have acute promyelocytic leukemia (APL) based on morphology, immunophenotype, molecular assay, or karyotype.
2. Participant has favorable risk cytogenetics
3. Participants with AML who may receive fms-like tyrosine kinase 3 (FLT3) inhibitor directed therapy.
4. Participant has or is suspected of having active central nervous system (CNS) involvement.
5. Participant has an active, uncontrolled infection except participants with infection under active treatment and controlled with antibiotics, antifungals, or antivirals are eligible.
6. Participant with prior autologous hematopoietic stem cell transplant (HSCT) who, in the investigator's judgment, have not fully recovered from the effects of the last transplant (eg, transplant related side effects).
7. Participant had prior allogeneic HSCT with either standard or reduced intensity conditioning ≤ 6 months prior to dosing.
8. Participants on systemic immunosuppressive therapy post HSCT at the time of screening, or with clinically significant graft-versus-host disease (GVHD). The use of topical steroids for ongoing skin or ocular GVHD is permitted.
9. Participant has immediate life-threatening, severe complications of leukemia such as disseminated/uncontrolled infection, uncontrolled bleeding, pneumonia with hypoxia or shock, and/or disseminated intravascular coagulation. The participant should be afebrile for at least 72 hours.
10. Participants requiring treatment with strong or moderate CYP3A inhibitors/inducers.
11. Participant has ongoing treatment with chronic, therapeutic dosing of anticoagulants.
12. Participant has a history of concurrent secondary cancers requiring active, ongoing systemic treatment.
13. Participant has known human immunodeficiency virus (HIV) infection.
14. Participant has known chronic active hepatitis B virus (HBV) or hepatitis C virus (HCV).

    1. Participant who is seropositive due to HBV vaccination is eligible.
    2. Participant who has no active viral infection and is under adequate prophylaxis against HBV reactivation is eligible.
15. Participant is known to have dysphagia, short-gut syndrome, gastroparesis, or other conditions that limit the ingestion or gastrointestinal absorption of drugs administered orally.
16. Participant has impaired cardiac function or clinically significant cardiac diseases
17. Participant has consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges), or Star fruit within 3 days prior to first venetoclax dose through last dose of venetoclax.
18. Pregnant women are excluded from this study due to potential teratogenic and/or abortifacient effect of this therapy. Nursing mothers should stop breastfeeding in order to be eligible due to potential risk for Adverse Events (AEs) in a nursing infant.
19. Participant has had previous treatment with a lysine-specific demethylase 1A (LSD1) inhibitor.
20. Participant has any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the participant from participating in the study.
21. Participant has any condition including the presence of laboratory abnormalities, which places the participant at unacceptable risk if he/she were to participate in the study.
22. Participant has any condition that confounds the ability to interpret data from the study.
23. Participant received live COVID-19 vaccines within 30 days prior to initiation of study treatment
24. Participants currently in other interventional trials, including those for COVID-19, may not participate in BMS clinical trials until the protocol specific washout period is achieved. If a study participant has received an investigational COVID-19 vaccine or other investigational product designed to treat or prevent COVID-19 prior to screening, enrollment must be delayed until the biologic impact of the vaccine or investigational product is stabilized, as determined by discussion between the Investigator and the Medical Monitor.

    Part I only:
25. Participant had prior treatment with venetoclax for AML, either as monotherapy or in combination with other agents.

    Part II and Part III only:
26. Participant had prior treatment with hypomethylating agent (HMA) or chemotherapy for antecedent hematologic disorders. Prior treatment with hydroxyurea is permitted.
27. Participant has received systemic anticancer therapy (including investigational therapy), radiotherapy, or immunotherapy < 14 days or 5 half-lives, whichever is shorter, prior to the first dose of CC-90011.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2022-03-09 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) | From ICF signature until 28 days after last dose of CC- 90011 and all combination agents
  An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a participant during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the participant's health, including laboratory test values, regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a preexisting condition) should be considered an AE
Recommended Phase 2 dose (RP2D) | Up to approximately Cycle 1 (each cycle is 28 days)
  The RP2D will include evaluation of DLTs and MTD using NCI CTCAE criteria

SECONDARY OUTCOMES:
Complete remission (CR) Rate | Up to approximately 10 months
  Defined as the rate of achieving CR (as assessed by the Investigator and by programmatic outputs by the Sponsor)
Complete remission with partial hematologic recovery (CRh) Rate | Up to approximately 2 years
  Defined as the rate of achieving CRh (as assessed by the Investigator and by programmatic outputs by the Sponsor)
Overall response rate (ORR) | Up to approximately 2 years
  Defined as the rate of achieving CR/CRMRD-/CRi/PR/MLFS
Duration of response (CR) | Up to approximately 2 years
  Time from the first CR to the date of documented disease relapse or death, whichever is earlier.
Duration of response (CR/CRh) | Up to approximately 2 years
  Time from the first CR or CRh to the date of documented disease relapse or death, whichever is earlier.
Duration of response (CR/ CRMRD-/ CRi/ PR/MLFS) | Up to approximately 2 years
  Time from the first CR, CRMRD-, CRi, PR or MLFS to the date of documented disease relapse, progression, or death, whichever is earlier.
Event-free survival (EFs)_Part III Only | Up to approximately 2 years
  Time from study randomization to the date of treatment failure, relapse from CR or death from any cause, whichever comes first.
Overall survival (OS)_Part III Only | Up to approximately 2 years
  Time from study randomization to the date of death due to any cause.
Minimal residual disease (MRD) Response Rate_Part II and III only | Up to approximately 2 years
  The rate of having at least a one log reduction in disease burden or an MRD negative (10-3) test result.
Minimal residual disease (MRD) Conversion Rate_Part II and III Only | Up to approximately 2 years
  The rate of participants achieving MRD negativity (10-3) at any time on therapy.
Complete response with incomplete hematologic recovery (CRi) rate | Up to approximately 2 years
  Defined as the rate of achieving CRi (as assessed by the Investigator and by programmatic outputs by the Sponsor)
Duration of response (CR/CRi) | Up to approximately 2 years
  Time from the first CR or CRi to the date of documented disease relapse or death, whichever is earlier.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (17):
- United States (11):
  - Local Institution - 110, Duarte, California
  - Local Institution - 103, New Haven, Connecticut
  - Local Institution - 108, Miami, Florida
  - Local Institution - 111, Chicago, Illinois
  - Local Institution - 121, New York, New York
  - Local Institution - 118, Durham, North Carolina
  - Local Institution - 116, Cleveland, Ohio
  - Local Institution - 115, Columbus, Ohio
  - Local Institution - 104, Dallas, Texas
  - Local Institution - 101, Houston, Texas
  - Local Institution - 120, Seattle, Washington
- Local Institution - 202, Ghent, Belgium
- Local Institution - 401, Villejuif, France
- Spain (4):
  - Local Institution - 803, Barcelona
  - Local Institution - 800, Barcelona
  - Local Institution - 802, Madrid
  - Local Institution - 801, Seville

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm